CLINICAL TRIAL: NCT06926465
Title: EFFICACY OF ADDING TRUNK INTEGRATED KINETIC CHAIN EXERCISES TO CONVENTIONAL EXERCISE THERAPY PROGRAM IN SUBACROMIAL IMPINGEMENT SYNDROME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maria Romany Edwar Raoof, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: treating shoulder impingement
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Subacromial Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group A (conventional traetment) (Active Comparator): conventional treatment including (hot pack, Stretching of the pectoralis minor, Resisted shoulder external rotation , Prone Extension ,Prone Horizontal Abduction with External Rotation ,Side-lying Forward Flexion ,Posterior capsule stretch (sleeper stretch)
  Interventions: Other: Conventional treatment
- Experimental group B (Trunk integrated kinetic chain exercises ) (Other): This group will receive conventional treatment plus four trunk integrated kinetic chain exercises:
  1. Quadruped shoulder flexion
  2. Shoulder flexion with trunk rotation
  3. Shoulder external rotation from shoulder at 45° internal rotation and the elbow at 90° flexion with trunk rotation
  4. Shoulder external rotation from shoulder at 90° abduction and the elbow at 90° flexion while with trunk rotation
  Interventions: Other: Trunk integrated kinetic chain exercises

INTERVENTIONS:
Other: Conventional treatment — conventional treatment including (hot pack, Stretching of the pectoralis minor, Resisted shoulder external rotation , Prone Extension ,Prone Horizontal Abduction with External Rotation ,Side-lying Forward Flexion ,Posterior capsule stretch (sleeper stretch)
  Arms: control group A (conventional traetment)
Other: Trunk integrated kinetic chain exercises — This group will receive conventional treatment plus four trunk integrated kinetic chain exercises:
  1. Quadruped shoulder flexion
  2. Shoulder flexion with trunk rotation
  3. Shoulder external rotation from shoulder at 45° internal rotation and the elbow at 90° flexion with trunk rotation
  4. Shoulder external rotation from shoulder at 90° abduction and the elbow at 90° flexion while with trunk rotation
  Arms: Experimental group B (Trunk integrated kinetic chain exercises )

SUMMARY:
The purpose of this study will be to investigate the effect of adding trunk integrated kinetic chain exercises to conventional exercise program on shoulder pain, function, isometric muscle strength, shoulder ROM and scapular orientation in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
Shoulder pain is the third most common musculoskeletal condition, affecting 67% of the general population . Shoulder impingement syndrome (SIS) is one of the most prevalent causes of shoulder pain, which is characterized by the compression of the rotator cuff and the subacromial bursa under subacromial space. Shoulder impingement syndrome is accounting for 44% to 65% of all shoulder complaints, with an estimated prevalence of 7% to 34%. In as many as 65% of SIS cases, shoulder pain is located in the anterolateral acromial region that may also spread to the lateral mid-humerus is the classic SIS symptom with a general decline in muscle strength.

New perspective for assessment and treatment of SIS is concentrating on movement-related mechanisms or biomechanical triggering factors. Exercises are effective at an early stage of SIS, which usually refers to stage I or early stage II according to Near's classification , such as training of the periscapular muscles (pectoralis minor, trapezius, serratus, and rhomboids) and strengthening of the rotator cuff (supraspinatus, infraspinatus, teres minor, and subscapularis), which acts as the shoulder joint stabilizers using concentric and eccentric exercises for the dynamic humeral centering effect and reduction of shoulder pain.). However, the best treatment strategy remains unknown If conservative treatment is failed operative treatment should be considered.

The scapula and glenohumeral joints are critical in allowing energy transfer from the trunk to lower limbs. According to Kibler et al, 1995, a 20% drop in kinetic energy transferred from the hip and trunk to the arm needs a 34% increase in shoulder rotational velocity to create the same amount of force to the hand. Deficiencies in the strength and mobility in these areas can have a negative impact on shoulder kinematics, increasing the risk of shoulder and elbow injury.

The defect at any link in the kinetic chain (Kc) will affect force transfer to subsequent segments and other components in the chain need to contribute more to compensate for the energy loss and this is explaining the risk factor for shoulder injury and pain. Recently, physical therapists typically recommend including lower extremity and trunk movements into shoulder rehabilitation protocols to maximize effective energy transfer throughout the entire KC. However, the importance of a KC approach over an isolated local shoulder treatment protocol during shoulder rehabilitation is not fully understood.

Previous studies investigated the efficacy of integrating the KC exercises into shoulder rehabilitation exercises and showed improvement of axio-scapular muscle recruitment, lower trapezius muscle ratios, and decrease the demands on the rotator cuff muscles.

A study examined EMG activity of the serratus anterior (SA) and lower trapezius (LT) during arm elevation this study and showed the highest activity of the SA, LT and Posterior Deltoid compared with the free-motion exercises. The quadruped shoulder flexion (QSF) is a form of KC ex in this study.

An EMG study analysis compared the muscle activation pattern of four Kc exercises to three conventional exercises the results showed that KC exercises resulted in the highest activation of all exercises. And this study is made on healthy subjects; if the examination is done on patients with shoulder pain the results may give different trends.

Furthermore, Yamauchi et al, (2015) investigated the effect of ipsilateral trunk rotation during shoulder exercises on the scapula. All Scaption, external rotations (ERs), and trunk rotation reported an increase of scapular ER or posterior tilt and LT activation. Retraction with 90° and 145° of shoulder abduction with trunk rotation considerably reduced UT activation and the UT/MT and UT/LT ratios. Therefore, the study findings imply that integrated trunk rotation KC ex adopted in this study may be useful in individuals with decreased (LT) activity and excessive (UT) activation or in cases where there is a diminished scapular ER or posterior tilt.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients complaining of subacromial impingement syndrome . 2) Age 20-¬45 years old . 3) If they had at least three of the following 6 criteria: "Neer sign" positive, "Hawkins sign" positive, " Painful active shoulder elevation in scapular plane, painful rotary cuff tendon palpation," painful resisted isometric abduction " history of pain related to C5 dermatome.

  4) A 20 percent or higher score of SPADI (Shoulder Pain and Disability Index) baseline 5) Level of pain (at least 2/10 on VAS) 6) Patient with Body mass index (BMI) with 18 to 29.5 Kg/m2

Exclusion Criteria:

1. Prior history of cervical radiculopathy symptoms, frozen shoulder
2. Neurological disorders, inflammatory disorders
3. Complete RC tear and any previous surgery to the affected shoulder
4. Infections or tumors

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Digital Goniometer | at baseline, to the end of treatment at 4 weeks
  to measure the full shoulder ROM using digital goniometer device in degrees
Hand held Dynamometer | at baseline, to the end of treatment at 4 weeks
  to measure shoulder and scapular muscle strength using hand held dynamometer , in newton

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic at faculty of physical therapy - Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lluch-Girbes E, Requejo-Salinas N, Fernandez-Matias R, Revert E, Vila Mejias M, Rezende Camargo P, Jaggi A, Sciascia A, Horsley I, Pontillo M, Gibson J, Richardson E, Johansson F, Maenhout A, Oliver GD, Turgut E, Jayaraman C, Duzgun I, Borms D, Ellenbecker T, Cools A. Kinetic chain revisited: consensus expert opinion on terminology, clinical reasoning, examination, and treatment in people with shoulder pain. J Shoulder Elbow Surg. 2023 Aug;32(8):e415-e428. doi: 10.1016/j.jse.2023.01.018. Epub 2023 Feb 15. PMID 36796714
- [Background] Lopes AD, Timmons MK, Grover M, Ciconelli RM, Michener LA. Visual scapular dyskinesis: kinematics and muscle activity alterations in patients with subacromial impingement syndrome. Arch Phys Med Rehabil. 2015 Feb;96(2):298-306. doi: 10.1016/j.apmr.2014.09.029. Epub 2014 Oct 15. PMID 25449194
- [Background] Maciel NFB, de Oliveira Sousa C. Motor alterations in the kinetic chain in individuals with chronic shoulder pain. Gait Posture. 2022 Mar;93:183-190. doi: 10.1016/j.gaitpost.2022.02.012. Epub 2022 Feb 13. PMID 35182984
- [Background] Mejia-Hernandez K, Chang A, Eardley-Harris N, Jaarsma R, Gill TK, McLean JM. Smartphone applications for the evaluation of pathologic shoulder range of motion and shoulder scores-a comparative study. JSES Open Access. 2018 Mar 13;2(1):109-114. doi: 10.1016/j.jses.2017.10.001. eCollection 2018 Mar. PMID 30675577
- [Background] Michener LA, McClure PW, Karduna AR. Anatomical and biomechanical mechanisms of subacromial impingement syndrome. Clin Biomech (Bristol). 2003 Jun;18(5):369-79. doi: 10.1016/s0268-0033(03)00047-0. PMID 12763431
- [Background] Michener LA, Boardman ND, Pidcoe PE, Frith AM. Scapular muscle tests in subjects with shoulder pain and functional loss: reliability and construct validity. Phys Ther. 2005 Nov;85(11):1128-38. PMID 16253043
- [Background] Nagai K, Tateuchi H, Takashima S, Miyasaka J, Hasegawa S, Arai R, Tsuboyama T, Ichihashi N. Effects of trunk rotation on scapular kinematics and muscle activity during humeral elevation. J Electromyogr Kinesiol. 2013 Jun;23(3):679-87. doi: 10.1016/j.jelekin.2013.01.012. Epub 2013 Feb 18. PMID 23428332
- [Background] Nakamura Y, Tsuruike M, Ellenbecker TS. Electromyographic Activity of Scapular Muscle Control in Free-Motion Exercise. J Athl Train. 2016 Mar;51(3):195-204. doi: 10.4085/1062-6050-51.4.10. Epub 2016 Mar 17. PMID 26986055
- [Background] Nazari G, MacDermid JC, Bryant D, Athwal GS. The effectiveness of surgical vs conservative interventions on pain and function in patients with shoulder impingement syndrome. A systematic review and meta-analysis. PLoS One. 2019 May 29;14(5):e0216961. doi: 10.1371/journal.pone.0216961. eCollection 2019. PMID 31141546
- [Background] Nijs J, Roussel N, Vermeulen K, Souvereyns G. Scapular positioning in patients with shoulder pain: a study examining the reliability and clinical importance of 3 clinical tests. Arch Phys Med Rehabil. 2005 Jul;86(7):1349-55. doi: 10.1016/j.apmr.2005.03.021. PMID 16003663
- [Background] Oliver GD, Plummer HA, Gascon SS. Electromyographic Analysis of Traditional and Kinetic Chain Exercises for Dynamic Shoulder Movements. J Strength Cond Res. 2016 Nov;30(11):3146-3154. doi: 10.1519/JSC.0000000000001389. PMID 26937768
- [Background] Phadke V, Camargo P, Ludewig P. Scapular and rotator cuff muscle activity during arm elevation: A review of normal function and alterations with shoulder impingement. Rev Bras Fisioter. 2009 Feb 1;13(1):1-9. doi: 10.1590/S1413-35552009005000012. PMID 20411160
- [Background] Phongamwong C, Choosakde A. Reliability and validity of the Thai version of the Shoulder Pain and Disability Index (Thai SPADI). Health Qual Life Outcomes. 2015 Sep 4;13:136. doi: 10.1186/s12955-015-0333-2. PMID 26337915
- [Background] Pieters L, Lewis J, Kuppens K, Jochems J, Bruijstens T, Joossens L, Struyf F. An Update of Systematic Reviews Examining the Effectiveness of Conservative Physical Therapy Interventions for Subacromial Shoulder Pain. J Orthop Sports Phys Ther. 2020 Mar;50(3):131-141. doi: 10.2519/jospt.2020.8498. Epub 2019 Nov 15. PMID 31726927
- [Background] Richardson E, Lewis JS, Gibson J, Morgan C, Halaki M, Ginn K, Yeowell G. Role of the kinetic chain in shoulder rehabilitation: does incorporating the trunk and lower limb into shoulder exercise regimes influence shoulder muscle recruitment patterns? Systematic review of electromyography studies. BMJ Open Sport Exerc Med. 2020 Apr 22;6(1):e000683. doi: 10.1136/bmjsem-2019-000683. eCollection 2020. PMID 32405430
- [Background] Rosa DP, Borstad JD, Pogetti LS, Camargo PR. Effects of a stretching protocol for the pectoralis minor on muscle length, function, and scapular kinematics in individuals with and without shoulder pain. J Hand Ther. 2017 Jan-Mar;30(1):20-29. doi: 10.1016/j.jht.2016.06.006. Epub 2016 Oct 18. PMID 27769843
- [Background] Rosa DP, Borstad JD, Ferreira JK, Gava V, Santos RV, Camargo PR. Comparison of specific and non-specific treatment approaches for individuals with posterior capsule tightness and shoulder impingement symptoms: A randomized controlled trial. Braz J Phys Ther. 2021 Sep-Oct;25(5):648-658. doi: 10.1016/j.bjpt.2021.04.003. Epub 2021 May 4. PMID 34001426
- [Background] Savoie A, Mercier C, Desmeules F, Fremont P, Roy JS. Effects of a movement training oriented rehabilitation program on symptoms, functional limitations and acromiohumeral distance in individuals with subacromial pain syndrome. Man Ther. 2015 Oct;20(5):703-8. doi: 10.1016/j.math.2015.04.004. Epub 2015 Apr 14. PMID 25907145
- [Background] Schydlowsky P, Szkudlarek M, Madsen OR. Comprehensive supervised heavy training program versus home training regimen in patients with subacromial impingement syndrome: a randomized trial. BMC Musculoskelet Disord. 2022 Jan 15;23(1):52. doi: 10.1186/s12891-021-04969-0. PMID 35033043
- [Background] Shadmehr A, Bagheri H, Ansari NN, Sarafraz H. The reliability measurements of lateral scapular slide test at three different degrees of shoulder joint abduction. Br J Sports Med. 2010 Mar;44(4):289-93. doi: 10.1136/bjsm.2008.050872. Epub 2008 Sep 23. PMID 18812417
- [Background] Shimizu H, Saito T, Kouno C, Shimoura K, Kawabe R, Shinohara Y, Mukaiyama K, Changyu C, Kato M, Nagai-Tanima M, Aoyama T. Validity and reliability of a smartphone application for self-measurement of active shoulder range of motion in a standing position among healthy adults. JSES Int. 2022 May 5;6(4):655-659. doi: 10.1016/j.jseint.2022.04.005. eCollection 2022 Jul. PMID 35813133
- [Background] Shin SH, Ro du H, Lee OS, Oh JH, Kim SH. Within-day reliability of shoulder range of motion measurement with a smartphone. Man Ther. 2012 Aug;17(4):298-304. doi: 10.1016/j.math.2012.02.010. Epub 2012 Mar 13. PMID 22421186
- [Background] Shire AR, Staehr TAB, Overby JB, Bastholm Dahl M, Sandell Jacobsen J, Hoyrup Christiansen D. Specific or general exercise strategy for subacromial impingement syndrome-does it matter? A systematic literature review and meta analysis. BMC Musculoskelet Disord. 2017 Apr 17;18(1):158. doi: 10.1186/s12891-017-1518-0. PMID 28416022
- [Background] Struyf F, Nijs J, Mottram S, Roussel NA, Cools AM, Meeusen R. Clinical assessment of the scapula: a review of the literature. Br J Sports Med. 2014 Jun;48(11):883-90. doi: 10.1136/bjsports-2012-091059. Epub 2012 Jul 21. PMID 22821720
- [Background] Turgut E, Duzgun I, Baltaci G. Effects of Scapular Stabilization Exercise Training on Scapular Kinematics, Disability, and Pain in Subacromial Impingement: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Oct;98(10):1915-1923.e3. doi: 10.1016/j.apmr.2017.05.023. Epub 2017 Jun 24. PMID 28652066
- [Background] Tsuruike M, Ellenbecker TS. Serratus anterior and lower trapezius muscle activities during multi-joint isotonic scapular exercises and isometric contractions. J Athl Train. 2015 Feb;50(2):199-210. doi: 10.4085/1062-6050-49.3.80. Epub 2014 Nov 14. PMID 25689561
- [Background] Yamauchi T, Hasegawa S, Matsumura A, Nakamura M, Ibuki S, Ichihashi N. The effect of trunk rotation during shoulder exercises on the activity of the scapular muscle and scapular kinematics. J Shoulder Elbow Surg. 2015 Jun;24(6):955-64. doi: 10.1016/j.jse.2014.10.010. Epub 2015 Jan 1. PMID 25556806
- [Background] Yuan X, Lowder R, Aviles-Wetherell K, Skroce C, Yao KV, Soo Hoo J. Reliability of point-of-care shoulder ultrasound measurements for subacromial impingement in asymptomatic participants. Front Rehabil Sci. 2022 Aug 17;3:964613. doi: 10.3389/fresc.2022.964613. eCollection 2022. PMID 36189022